CLINICAL TRIAL: NCT03868969
Title: Clinical Efficacy of Fosfomycin Trometamol Per os in the Treatment of Documented Male Urinary Tract Infections With ESBL-producing Enterobacteriaceae With ESBL Producing Enterobacteriaceae and Resistance Associated With Fluoroquinolones and Cotrimoxazole (FOSF'HOM)
Acronym: FOSF'HOM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: API/2017/90
Record Dates: First submitted 2019-03-04; First posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-02

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fosfomycin (Experimental): Fosomycin tromethamine, one sachet for 21 days
  Interventions: Drug: Fosfomycin Oral Suspension

INTERVENTIONS:
Drug: Fosfomycin Oral Suspension — Man with urinary tract infections with BLSE enterobacteriaceae will be treated by fosfomycin 1 packet by day for 21 days

SUMMARY:
The aim of the study was to evaluate the clinical and microbiological efficacy of fosfomycin trometamol (FT) per os in the treatment of documented male urinary tract infections with ESBL-producing enterobacteriaceae

ELIGIBILITY:
Inclusion Criteria:

* clinical suspicion of urinary tract infection (UTI) defined by the presence of at least one of these signs: fever > 38°C and/or sus-pubic pain and/or dysuria and/or pollakiuria and/or urinary burns and/or macroscopic hematuria and/or acute urinary retention and/or pain with the rectal examination and/or confusion
* And urinary analysis with leukocyturia > 10 / mm3, bacteriuria > 10^3 CFU/mL with ESBL producing enterobacteriaceae and resistance associated with fluoroquinolones (FQ) and cotrimoxazole (CTX) but sensitive to fosfomycin.

Exclusion Criteria:

* allergy to fosfomycin and/or trometamol
* Presence of material in the urinary tract
* Severe immunosuppression
* Chronic prostatitis
* Prostate abscess
* Acute pyelonephritis
* Hemodynamic instability
* Chronic renal failure (clearance <60 mL/min)
* Prior antibiotic therapy, with an antibiotic sensitive on the antibiotic susceptibility test except: amoxicillin - clavulanic acid, cefixime, nitrofurantoin.
* Co-treatment with metoclopramide

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients with no signs of urinary tract infection | 28 days
  Number of patients with no signs of urinary tract infection

SECONDARY OUTCOMES:
Number of patients with persistence of clinical signs of urinary tract infection | 3 days
  Number of patients with persistence of clinical signs of urinary tract infection
Number of patients with reoccurrence of clinical signs of urinary tract infection and positive urinary analysis | 3 months
  Number of patients with reoccurrence of clinical signs of urinary tract infection and positive urinary analysis
Number of patients with digestive, cutaneous disturbance | 28 days
  Number of patients with digestive, cutaneous disturbance

CONTACTS AND LOCATIONS:
Locations (1):
- BOUILLER, Besançon, France